CLINICAL TRIAL: NCT06202521
Title: Evaluation of the Safety and Efficacy of Silmitasertib (CX-4945) in Combination With Standard of Care (SOC) for Treating Patients With Community-Acquired Pneumonia (CAP) Associated With SARS-CoV-2 and Influenza Viral Infections
Brief Title: CX-4945 in Viral Community Acquired Pneumonia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial ended early in March 2025 due to changes in disease epidemiology, affecting patient availability and recruitment feasibility.
Sponsor: Senhwa Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CX-4945-011
Record Dates: First submitted 2024-01-01; First posted 2024-01-11 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Community-acquired Pneumonia; SARS-CoV-2 -Associated Pneumonia; Influenza With Pneumonia
Keywords: Covid-19; Influenza; Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia; COVID-19; Influenza, Human | interventions — silmitasertib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SARS-CoV-2 domain: CX-4945 (400 mg BID for 5 days) +SOC (Experimental): Notes: The SOC within the SARS-CoV-2 domain is defined as the medications in use at each respective site for the treatment of CAP related to SARS-CoV-2 infection.
  Interventions: Drug: CX-4945 (SARS-CoV-2 domain)
- SARS-CoV-2 domain: Placebo + SOC (Placebo Comparator): Notes: The SOC within the SARS-CoV-2 domain is defined as the medications in use at each respective site for the treatment of CAP related to SARS-CoV-2 infection.
  Interventions: Drug: Placebo (SARS-CoV-2 domain)
- Influenza virus domain: CX-4945 (400 mg BID for 5 days) +SOC (Experimental): Notes: The SOC within the influenza virus domain is defined as the medications in use at each respective site for the treatment of CAP related to influenza virus infection.
  Interventions: Drug: CX-4945 (Influenza virus domain)
- Influenza virus domain: Placebo + SOC (Placebo Comparator): Notes: The SOC within the influenza virus domain is defined as the medications in use at each respective site for the treatment of CAP related to influenza virus infection.
  Interventions: Drug: Placebo (Influenza virus domain)

INTERVENTIONS:
Drug: CX-4945 (SARS-CoV-2 domain) — CX-4945 will be administered at 400 mg BID for up to 5 days (Day 1 to Day 5) in addition to SOC.
  Other Names: Silmitasertib
  Arms: SARS-CoV-2 domain: CX-4945 (400 mg BID for 5 days) +SOC
Drug: Placebo (SARS-CoV-2 domain) — The dosage and frequency is the same as active drug.
  Arms: SARS-CoV-2 domain: Placebo + SOC
Drug: CX-4945 (Influenza virus domain) — CX-4945 will be administered at 400 mg BID for up to 5 days (Day 1 to Day 5) in addition to SOC.
  Other Names: Silmitasertib
  Arms: Influenza virus domain: CX-4945 (400 mg BID for 5 days) +SOC
Drug: Placebo (Influenza virus domain) — The dosage and frequency is the same as active drug.
  Arms: Influenza virus domain: Placebo + SOC

SUMMARY:
This is a Phase II, multi-center, double-blind, randomized, interventional study in approximately 120 subjects to evaluate clinical benefit of CX-4945 in adult outpatients with SARS-CoV-2 and influenza viral infection-associated pneumonia. The subjects will be recruited into two domains, including SARS-CoV-2 and influenza virus domains. The study will compare the efficacy of Standard of Care (SOC) combined with CX-4945 against SOC paired with a placebo, utilizing a 1:1 allocation ratio in each domain.

DETAILED DESCRIPTION:
Domain I: SARS-CoV-2 domain

* Arm 1: CX-4945 (400 mg BID for 5 days) +SOC
* Arm 2: Placebo + SOC

Domain II: Influenza virus domain

* Arm 3: CX-4945 (400 mg BID for 5 days) +SOC
* Arm 4: Placebo + SOC

Screening visit will collect health information and perform protocol specified tests to determine patients' eligibility. After screening visit, eligible subjects who fulfill all selection criteria for enrollment will be randomized into each of the arms. The CX-4945 will be administered at 400 mg BID for 5 days. Subjects will be followed up until Day 29.

ELIGIBILITY:
Inclusion Criteria

1. Not currently hospitalized
2. Males or females aged ≥ 18 years at the time of signing the informed consent form (ICF)
3. Patients diagnosed with viral pneumonia, as determined by the investigator, who exhibit any of the subsequent criteria: presence of respiratory symptoms or fever (ear temperature ≥ 38 °C, base of the tongue temperature ≥ 37.5 °C, or axillary temperature ≥ 37 °C)
4. With a pneumonia severity index (PSI) of risk class II or III
5. Oxygen saturation measured by pulse oximetry (SpO2) ≥ 94% on room air at sea level
6. Positive test for SARS-CoV-2 or influenza virus infection, confirmed by rapid diagnostic test (excluding cases where both SARS-CoV-2 and influenza virus are positive)
7. Confirmed lower respiratory tract infection by X-ray
8. At screening, subjects capable of childbearing must provide a negative serum or urine pregnancy test. These subjects must also commit to adhering to the study-specified contraceptive methods throughout the study duration

   Notes: Acceptable contraceptive methods include:
   * Established use of oral, injected or implanted hormonal methods of contraception
   * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
   * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps)
9. The participant (or legal representative) agrees and is able to adhere to study protocol-stated requirements, instructions, and restrictions in the investigator's judgement. Furthermore, the participant is capable of understanding and has signed the IRB-approved Informed Consent Form (ICF)
10. With at least two of the risk factors listed below: Age ≥ 50 years-old; cancer and a life expectancy of ≥ 6 months; HIV infection; immunocompromised patient; congestive heart failure (CHF), or coronary artery disease (CAD), or cardiomyopathies; chronic kidney disease (CKD); chronic liver disease; chronic lung disease; diabetes mellitus (DM); body mass index (BMI) > 25 kg/m2; asthma; cerebrovascular disease; cystic fibrosis; dementia; or current and former smoker

Exclusion Criteria

1. Subject received investigational treatment within 30 days prior to the study, or concurrent use of another investigational drug
2. Subject has a history of severe renal disease (required phosphate binders or dialysis)
3. Subject has chronic diarrhea, characterized by three or more loose stools daily for a minimum of four weeks
4. High likelihood of mortality within the next 48 hours, as assessed by the investigator
5. Subject showing signs of respiratory failure and mechanical ventilation is required
6. Subject with liver cirrhosis
7. Subject with hepatitis B and/or hepatitis C disease, unless the subject has an aspartate aminotransferase (AST) level ranging from 8 to 31 U/L and an alanine aminotransferase (ALT) level from 0 to 41 U/L
8. Known active tuberculosis
9. Current documented bacterial infection
10. Subject has a documented anaphylactic reaction, regardless of cause
11. Subject who has taken an antiviral agent against respiratory viral infection for a continuous duration of more than 24 hours before screening
12. Subject is with active gastrointestinal diseases including gastritis, ulcerative colitis, Crohn's disease, or hemorrhagic coloproctitis
13. Subjects received warfarin within 14 days prior to screening or intend to during the screening or treatment phase
14. History of allergic reactions to any of the ingredients or components used in the manufacture of CX-4945
15. Women who are pregnant or breastfeeding, or planning pregnancy during the study

    Note: Men and women of reproductive potential must commit to effective contraception methods or abstinence during the study. Any resulting pregnancies or suspected pregnancies must be reported to the treating physician immediately.
16. ALT or AST levels > 5 times upper limit of normal (ULN)
17. eGFR <30 mL/min/1.73m2 (calculated by the MDRD formula)
18. Absolute neutrophil count (ANC) <1000/μL
19. Have received treatment with a SARS-CoV-2 specific monoclonal antibody
20. Have received convalescent COVID-19 plasma treatment
21. Concurrent use of baricitinib
22. Any physical findings or illness history that may compromise study results or increase patient risk, as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Huang, M.D., Study Chair — Senhwa Biosciences
Locations (7):
- Taiwan (7):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Cancer Center, National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from individuals diagnosed with Community-Acquired Pneumonia (CAP) associated with SARS-CoV-2 and influenza viral infections at seven sites across Taiwan between February 2024 and March 2025. The first participant was enrolled on March 20, 2024, and the last on February 27, 2025.
Pre-assignment Details: Of the 45 enrolled participants, 44 met inclusion criteria and were randomized.
Groups:
- SARS-CoV-2 Domain: CX-4945 + SOC: Participants received Silmitasertib (CX-4945) 400 mg capsules orally twice a day for 5 days. Participants received Standard of Care (SOC) as assigned by the investigator.
  Notes: The SOC within the SARS-CoV-2 domain is defined as the medications in use at each respective site for the treatment of CAP related to SARS-CoV-2 infection.
- SARS-CoV-2 Domain: Placebo + SOC: Participants received Placebo capsules orally twice a day for 5 days. Participants received Standard of Care (SOC) as assigned by the investigator.
  Notes: The SOC within the SARS-CoV-2 domain is defined as the medications in use at each respective site for the treatment of CAP related to SARS-CoV-2 infection.
- Influenza Virus Domain: CX-4945 + SOC: Participants received Silmitasertib (CX-4945) 400 mg capsules orally twice a day for 5 days. Participants received Standard of Care (SOC) as assigned by the investigator.
  Notes: The SOC within the influenza virus domain is defined as the medications in use at each respective site for the treatment of CAP related to influenza virus infection.
- Influenza Virus Domain: Placebo + SOC: Participants received Placebo capsules orally twice a day for 5 days. Participants received Standard of Care (SOC) as assigned by the investigator.
  Notes: The SOC within the influenza virus domain is defined as the medications in use at each respective site for the treatment of CAP related to influenza virus infection.
Period: Overall Study
Arm/Group | SARS-CoV-2 Domain: CX-4945 + SOC | SARS-CoV-2 Domain: Placebo + SOC | Influenza Virus Domain: CX-4945 + SOC | Influenza Virus Domain: Placebo + SOC
Started | 15 | 15 | 7 | 7
Completed | 15 | 14 | 6 | 6
Not Completed | 0 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population is defined as all randomized subjects who received at least one dose of Silmitasertib (CX-4945) or placebo. This population was used as the primary analysis population for efficacy endpoints and the analysis population for baseline data, safety and exploratory endpoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | SARS-CoV-2 Domain: CX-4945 + SOC | SARS-CoV-2 Domain: Placebo + SOC | Influenza Virus Domain: CX-4945 + SOC | Influenza Virus Domain: Placebo + SOC | Total
Number analyzed (Participants) | 15 | 15 | 7 | 7 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.3 (11.88) | 47.4 (11.04) | 48.6 (13.35) | 49.0 (14.33) | 47.5 (11.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 2 | 4 | 23
  Male | 6 | 7 | 5 | 3 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 15 | 7 | 7 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Requiring Hospitalization, Including Emergency Room Visits, or Resulting in Death Due to Progression of CAP Related to SARS-CoV-2 or Influenza.
Description: To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared to placebo plus SOC, in preventing the progression of CAP associated with SARS-CoV-2 and influenza virus infection
Time Frame: Day 1 to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 15 | 15 | 7 | 7
Participants | 0 | 0 | 0 | 0

2. Secondary Outcome: The Percentage of Subjects With All Cause Hospitalization, Emergency Room Visits, or Death During Study Period.
Description: To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition
Time Frame: Day 1 to Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 15 | 15 | 7 | 7
Participants | 0 | 1 | 1 | 0

3. Secondary Outcome: The Percentage of Subjects With Improved Pulmonary X-ray Findings for Pneumonia, Relative to Baseline or Showing a Return to Normalcy
Description: To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition.
  Note: Visit 3 and its associated efficacy/safety assessments were scheduled for Day 5 in protocol version 1.0 and for Day 7 since protocol version 2.0.
Time Frame: Baseline to Day 5/7
Population: The participant who has completed Day 5/7, Day 15 or Day 29 is eligible for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 15 | 15 | 7 | 7
Participants
  Day 5/7: number analyzed (Participants) | 15 | 15 | 7 | 6
  Day 5/7: Worsen | 1 | 1 | 1 | 0
  Day 5/7: No change | 1 | 1 | 3 | 0
  Day 5/7: Improved | 8 | 7 | 1 | 5
  Day 5/7: Normal | 5 | 6 | 2 | 1
  Day 15: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 15: Worsen | 0 | 0 | 0 | 0
  Day 15: No change | 1 | 0 | 0 | 0
  Day 15: Improved | 5 | 5 | 3 | 2
  Day 15: Normal | 9 | 9 | 3 | 4
  Day 29: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 29: Worsen | 0 | 0 | 0 | 0
  Day 29: No change | 0 | 0 | 0 | 0
  Day 29: Improved | 1 | 0 | 2 | 0
  Day 29: Normal | 14 | 14 | 4 | 6

4. Secondary Outcome: The Symptom Resolution for Fever is Defined as Body Temperature Lower Than the Following Definition for 24 Hours (Ear Temperature < 38 °C, Base of the Tongue Temperature < 37.5 °C, or Axillary Temperature < 37 °C)
Description: Time to Symptom Resolution for Fever [days]. The symptom resolution for fever is defined as body temperature lower than the following definition (ear temperature < 38 °C, base of the tongue temperature < 37.5 °C, or axillary temperature < 37 °C) Note: Visit 3 and its associated efficacy/safety assessments were scheduled for Day 5 in protocol version 1.0 and for Day 7 since protocol version 2.0.
Time Frame: Day 1 to Day 5/7
Population: The participants were observed to have fever at baseline.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 1 | 1 | 3 | 3
days | 1.8 [NA to NA] — only 1 participant Analyzed | 1.2 [NA to NA] — only 1 participant Analyzed | 1.8 [1.20 to NA] — insufficient number of participants with events | 1.7 [1.50 to NA] — insufficient number of participants with events

5. Secondary Outcome: Change From Baseline in SpO2/FiO2 Ratio
Description: To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition Note: Visit 3 and its associated efficacy/safety assessments were scheduled for Day 5 in protocol version 1.0 and for Day 7 since protocol version 2.0.
Time Frame: Day 1 to Day 5/7, 15, and 29
Population: The participant who has completed Day 5/7, Day 15 or Day 29 is eligible for analysis.
Measure: Mean (Standard Deviation); unit: ratio change
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 15 | 15 | 7 | 7
ratio change
  Day 5/7 | 0.95 (3.689) | 0.63 (4.359) | 2.04 (4.647) | 0.68 (5.091)
  Day 15: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 15 | 0.95 (2.670) | 1.36 (4.736) | 3.17 (6.506) | 1.59 (3.888)
  Day 29: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 29 | 1.59 (3.446) | 1.70 (6.083) | 4.76 (3.012) | 2.38 (5.832)

6. Secondary Outcome: The Percentage of Subjects Exhibiting Disease Progression in Health Status Disease Progression is Defined as an Increase of Score on the National Institute of Allergy and Infectious Diseases (NIAID) 8-point Ordinal Scale
Description: To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition.
  NIAID 8-point ordinal scale range: 1-8, with higher scores indicating a worse condition.
  Note: Visit 3 and its associated efficacy/safety assessments were scheduled for Day 5 in protocol version 1.0 and for Day 7 since protocol version 2.0.
Time Frame: Day 1 to Day 5/7, 15, and 29
Population: The participant who has completed Day 5/7, Day 15 or Day 29 is eligible for analysis.
  Calculate the percentage of subjects whose health condition has progressed.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 15 | 15 | 7 | 7
Participants
  Day 5/7 | 0 | 0 | 0 | 0
  Day 15: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 15 | 0 | 0 | 1 | 0
  Day 29: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 29 | 0 | 0 | 0 | 0

7. Secondary Outcome: The Percentage of Subjects Exhibiting Health Improvement in Health Status Health Improvement is Defined as a Reduction of Score on the National Institute of Allergy and Infectious Diseases (NIAID) 8-point Ordinal Scale
Description: To evaluate the effect of intervention with Silmitasertib (CX-4945) in addition to SOC, compared with placebo plus SOC, in enhancing the subject's clinical condition NIAID 8-point ordinal scale range: 1-8, with higher scores indicating a worse condition.
  Note: Visit 3 and its associated efficacy/safety assessments were scheduled for Day 5 in protocol version 1.0 and for Day 7 since protocol version 2.0.
Time Frame: Day 1 to Day 5/7, 15, and 29
Population: The participant who has completed Day 5/7, Day 15 or Day 29 is eligible for analysis.
  Calculate the percentage of subjects whose health condition has improved.
Measure: Count of Participants; unit: Participants
Arm/Group | SARS-CoV-2 domain: CX-4945 + SOC | SARS-CoV-2 domain: Placebo + SOC | Influenza virus domain: CX-4945 + SOC | Influenza virus domain: Placebo + SOC
Number analyzed (Participants) | 15 | 15 | 7 | 7
Participants
  Day 5/7 | 2 | 1 | 2 | 1
  Day 15: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 15 | 4 | 2 | 2 | 1
  Day 29: number analyzed (Participants) | 15 | 14 | 6 | 6
  Day 29 | 5 | 2 | 2 | 1

ADVERSE EVENTS:
Time Frame: From randomization until end of follow-up, up to 32 days
Description: Adverse Events experienced by patients from randomization to Day 29 (± 3 days) (including vital signs, physical findings, clinical laboratory, and ECG results) as characterized by type, frequency, severity (as graded by Common Terminology Criteria for Adverse Events (CTCAE version 5.0), timing, seriousness, and relationship to study therapy.
Arm/Group | SARS-CoV-2 Domain: CX-4945 + SOC | SARS-CoV-2 Domain: Placebo + SOC | Influenza Virus Domain: CX-4945 + SOC | Influenza Virus Domain: Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 1/7 | 0/7
Other Adverse Events (participants affected / at risk) | 10/15 | 4/15 | 5/7 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SARS-CoV-2 Domain: CX-4945 + SOC (N=15) | SARS-CoV-2 Domain: Placebo + SOC (N=15) | Influenza Virus Domain: CX-4945 + SOC (N=7) | Influenza Virus Domain: Placebo + SOC (N=7)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced an SAE of Grade 3 unspecified bacterial pneumonia (unlikely related to the IP)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SARS-CoV-2 Domain: CX-4945 + SOC (N=15) | SARS-CoV-2 Domain: Placebo + SOC (N=15) | Influenza Virus Domain: CX-4945 + SOC (N=7) | Influenza Virus Domain: Placebo + SOC (N=7)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 1 (1) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suspected drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
This trial was terminated early on March 31, 2025 due to insufficient differentiation of the primary endpoint in addressing the unmet medical need, as well as recruitment difficulties caused by the end of the flu season.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2024-08-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT06202521/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT06202521/SAP_001.pdf